CLINICAL TRIAL: NCT03342508
Title: Outcomes Following Cesarean Delivery for Failure to Progress With Use of a Fetal Pillow
Brief Title: Fetal Pillow Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Julian N Robinson, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017P001986
Record Dates: First submitted 2017-09-08; First posted 2017-11-17 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Labor Complication
Keywords: Maternal outcomes; Neonatal Outcomes
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Each patient will have a Fetal Pillow inserted vaginally by the obstetrician after catheterization of the bladder (if it has not been previously performed). Once the Fetal Pillow is in place, the woman's legs will be placed flat on the operating table. The anesthesiologist will then inflate the Fetal Pillow if the patient has been randomized into the Fetal Pillow Inflated (FPI) group. In the Fetal Pillow Not Inflated (FPNI) group, the device will remain, not inflated, in the vagina. The obstetrician will therefore be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fetal Pillow Inflated (FPI) (Experimental): A Fetal Pillow will be inserted vaginally by the obstetrician after catheterization of the bladder (if it has not been previously performed). Once the Fetal Pillow is in place, the woman's legs will be placed flat on the operating table. The anesthesiologist will then inflate the Fetal Pillow. The obstetrician will not be aware to inflation of Fetal Pillow
  Cesarean delivery will then be performed
  The circulating nurse will deflate the Fetal Pillow following delivery. The obstetrician will remove the Fetal Pillow at the end of the procedure. The obstetrician will then fill out a survey regarding the delivery.
  Interventions: Device: Fetal Pillow
- Fetal Pillow Not Inflated (FPNI) (No Intervention): A Fetal Pillow will be inserted vaginally by the obstetrician after catheterization of the bladder (if it has not been previously performed). Once the Fetal Pillow is in place, the woman's legs will be placed flat on the operating table. The Fetal Pillow will not be inflated.
  Cesarean delivery will then be performed. The obstetrician will continue to be able to use conventional methods for delivery of a second stage arrest including hand from below and reverse breech extraction.
  The circulating nurse will deflate the Fetal Pillow following delivery. The obstetrician will remove the Fetal Pillow at the end of the procedure. The obstetrician will then fill out a survey regarding the delivery.

INTERVENTIONS:
Device: Fetal Pillow — see arm description
  Arms: Fetal Pillow Inflated (FPI)

SUMMARY:
The purpose of this study is to evaluate outcomes following cesarean delivery for failure to progress with the use of the Fetal Pillow. Our hypothesis is that time to delivery of the fetus is shorter with implementation of the Fetal Pillow.

DETAILED DESCRIPTION:
Women will be enrolled from the labor floor during their labor course when there is concern for cesarean section for failure to progress in the second stage of labor. These women may be approached if they have a prolonged labor course (before they reach full dilation), when they get to full dilation and start pushing, or following an unsuccessful operative delivery. All women who meet the inclusion criteria will be approached about participation in the study on labor and delivery. The process of informed consent will happen at that time on labor and delivery. All women will be enrolled by study staff or certain physicians at Brigham and Women's Hospital who have agreed to help consent patients for this study.

Once consent is obtained, the subjects will then be randomized 1:1 into two parallel groups, the Fetal Pillow Inflated (FPI) group and the Fetal Pillow Not Inflated (FPNI) group. A random number generator will allocate the groups in blocks of ten.

The Fetal Pillows used in the study have been donated by Safe Obstetrics Systems.

Each patient will have a Fetal Pillow inserted vaginally by the obstetrician after catheterization of the bladder (if it has not been previously performed). Once the Fetal Pillow is in place, the woman's legs will be placed flat on the operating table. The anesthesiologist will then inflate the Fetal Pillow if the patient has been randomized into the Fetal Pillow Inflated (FPI) group. In the Fetal Pillow Not Inflated (FPNI) group, the device will remain, not inflated, in the vagina. The obstetrician will therefore be blinded to the intervention. In the FPNI group the obstetrician will continue to be able to use conventional methods for delivery of a second stage arrest including hand from below and reverse breech extraction. The Fetal Pillow will be drained by the circulating nurse in the operating room following delivery with removal at the end of the procedure by the obstetrician.

ELIGIBILITY:
Inclusion Criteria:

* women age 18-50
* term pregnancy (37- 41 6/7 weeks)
* singleton gestation in cephalic presentation
* fully dilated
* both nulliparous and multiparous women
* both spontaneous labor and labor inductions

Exclusion Criteria:

* breech presentation
* presence of contraindication to vaginal delivery
* prior cesarean section
* presence of congenital anomalies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only women undergoing cesarean section are included
Enrollment: 60 (Actual)
Dates: Start 2018-01-13 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Uterine incision to delivery time | Assessed at time of delivery, delivery day (day 0)
  Time (in seconds) from hysterotomy to delivery

SECONDARY OUTCOMES:
Difficulty of Delivery of Fetal head | Assessed at time of delivery, delivery day (day 0)
  Score of difficulty of delivery 1-5 (1: very difficult, 5: very easy)
Uterine extension | Assessed at time of delivery, delivery day (day 0)
  Grading of extension 1-3
Composite Maternal Morbidity | Assessed both following delivery (day 0) and at end of study period (week 4)
  Blood loss, presence of blood transfusion, change in hematocrit from preop to postop day 1, temperature>100.4, ICU transfer, presence of Disseminated intravascular coagulation (DIC), readmission
Length of stay | Assessed at end of study period (week 4)
  Maternal Length of stay
Fetal Weight | Assessed at time of delivery, delivery day (day 0)
  Weight of fetus at time of birth
1 minute APGAR | Assessed at time of delivery, delivery day (day 0)
  Assessment of the 1 minute APGAR
5 minute APGAR | Assessed at time of delivery, delivery day (day 0)
  Assessment of the 5 minute APGAR
Composite Neonatal Morbidity | Assessed at end of study period (week 4)
  Need for intubation, fetal trauma
Neonatal Intensive Care Unit (NICU) Length of Stay | Assessed at end of study period (week 4)
  Length of stay in NICU
Provider Opinions | Assessed at end of study period (week 4)
  Willingness to recommend to others based on ease of placement and removal (1-5 point scale)

CONTACTS AND LOCATIONS:
Overall Officials: Julian N Robinson, MD, Principal Investigator — Brigham and Women's Hospital, Harvard Medical School, Boston MA
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mancuso MS, Rouse DJ. Cesarean delivery for abnormal labor. Clin Perinatol. 2008 Sep;35(3):479-90, ix. doi: 10.1016/j.clp.2008.06.004. PMID 18952016
- [Result] Myles TD, Santolaya J. Maternal and neonatal outcomes in patients with a prolonged second stage of labor. Obstet Gynecol. 2003 Jul;102(1):52-8. doi: 10.1016/s0029-7844(03)00400-9. PMID 12850607
- [Result] Safa H, Beckmann M. Comparison of maternal and neonatal outcomes from full-dilatation cesarean deliveries using the Fetal Pillow or hand-push method. Int J Gynaecol Obstet. 2016 Dec;135(3):281-284. doi: 10.1016/j.ijgo.2016.06.013. Epub 2016 Aug 24. PMID 27599604
- [Result] Seal SL, Dey A, Barman SC, Kamilya G, Mukherji J. Does elevating the fetal head prior to delivery using a fetal pillow reduce maternal and fetal complications in a full dilatation caesarean section? A prospective study with historical controls. J Obstet Gynaecol. 2014 Apr;34(3):241-4. doi: 10.3109/01443615.2013.844108. Epub 2014 Jan 31. PMID 24483234
- [Result] Seal SL, Dey A, Barman SC, Kamilya G, Mukherji J, Onwude JL. Randomized controlled trial of elevation of the fetal head with a fetal pillow during cesarean delivery at full cervical dilatation. Int J Gynaecol Obstet. 2016 May;133(2):178-82. doi: 10.1016/j.ijgo.2015.09.019. Epub 2016 Jan 15. PMID 26868074
- [Derived] Lassey SC, Little SE, Saadeh M, Patton N, Farber MK, Bateman BT, Robinson JN. Cephalic Elevation Device for Second-Stage Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2020 Apr;135(4):879-884. doi: 10.1097/AOG.0000000000003746. PMID 32168216